CLINICAL TRIAL: NCT05899036
Title: PULSE-C: Early Feasibility Study of RapidPulseTM Aspiration System as Frontline Approach for Patients With Acute Ischemic Stroke Due to Large Vessel Occlusions
Brief Title: Early Feasibility Study of RapidPulseTM Aspiration System for Patients With Acute Ischemic Stroke
Acronym: PULSE-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RapidPulse, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0003
Record Dates: First submitted 2023-05-16; First posted 2023-06-12 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke; Stroke; Large Vessel Occlusion; Mechanical Thrombectomy
Keywords: Stroke; Mechanical Thrombectomy
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Thrombectomy

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, open-label, single-arm study to assess the initial technical (performance), effectiveness, and safety of the RapidPulseTM Aspiration System. As such, no formal statistical hypothesis will be tested in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Each subject will undergo baseline evaluation for acute ischemic stroke due to large vessel occlusion, per standard of care and undergo mechanical thrombectomy procedure, aspiration to remove the thrombus in the neuro-vasculature using the RapidPulseTM Aspiration System.
  Interventions: Device: RapidPulseTM Aspiration System

INTERVENTIONS:
Device: RapidPulseTM Aspiration System — The RapidPulseTM Aspiration System is designed to remove occlusive thrombus from the cerebral vasculature using pulsatile aspiration. The system is comprised of a sterile one-time use 071 catheter, a sterile one-time use tubing set and a multiuse aspiration pump console.
  Other Names: Aspiration Thrombectomy; Thrombectomy

SUMMARY:
The goal of this clinical trial is to assess the initial safety and performance of the RapidPulseTM Aspiration System in patients experiencing acute ischemic stroke within 24 hours since the onset of stroke symptoms, or last known normal. Subject will undergo mechanical thrombectomy (a procedure to remove a clot in the brain which is preventing blood flow), with the RapidPulseTM Aspiration System. Participating in the trial is for 5-7 days or hospital discharge (whichever is earlier).

DETAILED DESCRIPTION:
The purpose of this prospective, multi-center, open label study of the RapidPulseTM Aspiration System is to assess the initial technical (performance), effectiveness and safety of the RapidPulseTM Aspiration System as frontline approach for patients with acute ischemic stroke due to large vessel occlusions identified within 24 hours of symptom onset (or last seen normal). The target sample size is 10 evaluable subjects with a maximum of 50 subjects. Subjects will undergo mechanical thrombectomy procedure and will have postoperative assessments completed at 24 hours and on Day 5-7 or upon hospital discharge. The primary endpoint is first pass reperfusion effect (FPE) as defined by mTICI ≥ 2c after one reperfusion attempt.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke with symptom onset (or last seen normal) within 24 hours.
* CTA, MRA or DSA demonstrating anterior large vessel occlusion involving the intracranial ICA, MCA M1 or M2 segments, basilar or vertebral artery
* Target occlusion can be accessed by the RapidPulseTM 071 aspiration catheter assessed at the time of the index procedure. Enrollment will be defined by the successful navigation of the RapidPulseTM 071 aspiration catheter into the occlusion site.

Exclusion Criteria:

* Known or suspected ICAD
* Tandem occlusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-03-23 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
First Pass Reperfusion Effect (FPE) | Intra-procedural
  The number of subjects with mTICI ≥ 2c after one reperfusion attempt

OTHER OUTCOMES:
Frontline technical success | Intra-procedural
  The number of subjects with mTICI ≥ 2b after the last pass with Study Device (no rescue therapy)
Final mTICI score | Intra-procedural
  The final mTICI score (0-3) for all subjects after all passes (including any rescue therapy)
Modified First Pass Reperfusion Effect (mFPE) | Intra-procedural
  The number of subjects with mTICI ≥ 2b after one device pass
Device-related and procedure-related adverse events | Intra and post procedural (up to Day 5-7 or discharge whichever occurs earlier)
  Including vessel injury, distal emboli, emboli in new territory (ENT) and vessel spasm

CONTACTS AND LOCATIONS:
Overall Officials: Raul G Nogueira, Study Chair — University of Pittsburgh Medical Center Stroke Institute
Locations (2):
- Hospital de Clinicas Facultad de Medicina-Universidad Nacional de Asunción, Asunción, Paraguay
- İstanbul Aydın Üniversitesi V.M Medical Park Florya Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No